CLINICAL TRIAL: NCT03581552
Title: A Pilot Study Examining Molecular and Clinical Effects of Aromatase Inhibitor Therapy on Skeletal Muscle Function in Early Stage Breast Cancer
Brief Title: Effects of Aromatase Inhibitor Therapy on Muscle Function
Status: Completed | Type: Observational
Sponsor: Tarah J Ballinger, MD (Other)
Responsible Party: Sponsor-Investigator, Tarah J Ballinger, MD, Assistant Professor of Clinical Medicine, Indiana University
Organization: Indiana University (Other)
Other Study IDs: IUSCC-0647
Record Dates: First submitted 2018-06-04; First posted 2018-07-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Breast Cancer Female
Keywords: Post Menopausal; ER positive; Aromatase Inhibitor Therapy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum blood samples will be collected to measure markers of bone turnover and to perform a serum TGF-β assay. Samples will be collected at baseline and within 14 days of day 168 of aromatase inhibitor (AI) treatment
  Skeletal muscle tissue will be collected and used to compare relative calstabin1 to RyR1 and RyR1 oxidation before and after exposure to aromatase inhibitor (AI) treatment. One sample will be stored for future research relating to aromatase inhibitor-induced muscle weakness including proteomic research. Four core needle samples will be taken from the quadriceps muscle at baseline and within 14 days of day 168 of AI treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot study designed to examine changes in muscle function after Aromatase Inhibitor (AI) therapy, at both the molecular and clinical level.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Post-menopausal
3. Diagnosis of ductal carcinoma in situ (DCIS) or stage I, II, or III ER positive breast cancer
4. Plan to initiate an AI per treating physician.
5. Completion of all primary therapy for breast cancer, including surgery, radiation, and chemotherapy (should be completed 14 days or more prior to obtaining the baseline muscle biopsy). Ongoing HER2 targeted therapy with trastuzumab and/or pertuzumab is allowed. Ongoing neratinib therapy is not allowed.
6. Body weight less than 350 lbs., as dictated by the weight limit for DXA (dual energy x-ray absorptiometry) scanner
7. Must be willing to undergo muscle biopsy at baseline and after 24 weeks of AI therapy
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 at the time of study enrollment
9. Informed consent and authorization of the release of health information must be obtained according to institutional guidelines

Exclusion Criteria:

1. Unwilling to co-enroll into the FIT core study
2. Diagnosis of severe osteopenia or osteoporosis, defined as a bone mineral density of ≥ 2.0 standard deviations below the young adult female reference mean (T score)
3. Diagnosis of other disorder affecting bone function or turnover, such as Paget's disease, renal osteodystrophy, parathyroid disorders, or vitamin D deficiency/osteomalacia
4. Prior history of non-traumatic, fragility bone fracture
5. Any muscle or neuromuscular disorder affecting muscle function, such as muscular dystrophy, myositis, or amyotrophic lateral sclerosis
6. Any condition precluding power protocol participation (i.e. exertion on a stationary bicycle), including: New York Heart Association (NYHA) class III or IV congestive heart failure, uncontrolled angina, myocardial infarction in the prior 12 months, orthopedic surgery in the previous 6 months or plans for orthopedic surgery during the study period, chronic uncontrolled pulmonary conditions such as uncontrolled asthma (symptoms > 2 days/week) or dyspnea requiring oxygen, symptomatic peripheral vascular disease, or any other comorbidity that would interfere with the ability to complete and comply with the protocol in the opinion of the investigator
7. Need for daily anticoagulation use
8. Allergy to local anesthetic
9. Locally recurrent or metastatic breast cancer a. History of prior treated malignancies, other than breast cancer, that are now stable, are in remission, and do not require active therapy, are acceptable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Post menopausal women with non metastatic breast cancer planning to initiate aromatase inhibitor therapy at the IU Simon Cancer Center oncology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Changes in calstabin1 binding to RyR1 channels in skeletal muscle | through day 168 of aromatase inhibitor therapy
  Changes in calstabin1 binding to RyR1 channels in skeletal muscle of breast cancer patients pre and post exposure to adjuvant aromatase inhibitor therapy

SECONDARY OUTCOMES:
Changes in ryanodine receptor/calcium release channel (RyR1) oxidation in skeletal muscle | through day 168 of aromatase inhibitor therapy
  To estimate changes in RyR1 oxidation in skeletal muscle of breast cancer patients, pre- and post- exposure to adjuvant aromatase inhibitor therapy
Relationship between changes in RyR1 biochemistry and measures of muscle function | through day 168 of aromatase inhibitor therapy
  To explore the relationship between changes in RyR1 biochemistry and measures of muscle function, including muscle power as measured by isokinetic dynamometry
Relationship between markers of bone turnover and changes in RyR1 biochemistry | through day 168 of aromatase inhibitor therapy
  To explore the relationship between markers of bone turnover and changes in RyR1 biochemistry (calstabin binding to RyR1)
Relationship between markers of bone turnover and changes in muscle function | through day 168 of aromatase inhibitor therapy
  To explore the relationship between markers of bone turnover and changes in muscle function in terms of muscle power assessed by isokinetic dynamometry
Characterize the timing of development of muscle dysfunction following initiation of aromatase inhibitor therapy | through day 168 of aromatase inhibitor therapy
  To better characterize the timing of development of muscle dysfunction following initiation of aromatase inhibitor therapy, in terms muscle power measured by isokinetic dynamometry
Feasibility of repeated muscle biopsies in patients with early stage breast cancer initiating aromatase inhibitor therapy | through day 168 of aromatase inhibitor therapy
  5. To describe the feasibility of repeated muscle biopsies in patients with early stage breast cancer initiating aromatase inhibitor therapy, in terms of rate of completion of baseline and follow up biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Tarah Ballinger, MD, Principal Investigator — Indiana University
Locations (1):
- IU Simon Cancer Center, Indianapolis, Indiana, United States